CLINICAL TRIAL: NCT06049537
Title: Studying Respiratory Infections and Colonisation in Children Using Daily Minimally-invasive Nasal Sampling
Acronym: SAMSAM
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Spaarne Gasthuis (Other)
Responsible Party: Principal Investigator, Simon P Jochems, PhD, assistant professor, Leiden University Medical Center
Other Study IDs: P21.067
Record Dates: First submitted 2023-08-31; First posted 2023-09-22 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Tract; Infection, Upper (Acute); Colonization, Asymptomatic
Keywords: Host-pathogen interactions; Minimally-invasive nasal sampling; Colonization/URT infections in children
MeSH Terms: conditions — Infections; Asymptomatic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples are collected at baseline (day 1) from children Nasopharyngeal swabs are collected at day 28 from children Saliva samples are collected at days 1, 14, 28 from children Nasosorption samples are collected from nose daily for entire study 28 days For a subset of parents of enrolled children, daily saliva samples are collected for 28 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young children: Children aged 1-5 years old attending school or day care. Follow-up for 28 days using minimally-invasive nasosorption sampling and questionnaires relating to symptoms.
  No intervention administered
- Parents: Parents of enrolled children, if it is a one-child family. Follow-up for 28 days using minimally-invasive saliva sampling.
  No intervention administered

SUMMARY:
Rationale: Respiratory tract infections (RTI) are a major cause of morbidity in young children in high- income countries and the major cause of mortality in developing countries. Causative bacteria and viruses are regular residents of the nasopharynx of asymptomatic individuals (colonization) and live there together with other presumed harmless commensals, without causing disease. These non-pathological infections/colonization episodes are important for transmission, intermediate step to disease and boost immune responses. The investigators recently validated the use of minimally-invasive nasal sampling methods that can be done at home for the study of host and microbial parameters in adults and children. In this study the investigators will focus on the daily microbial and immunological composition of the nasopharynx during health in relation to symptoms.

Primary objective: Associate acquisition of pneumococcal colonisation with levels of pre-existing polysaccharide specific memory B cells.

Secondary objectives include: Validate the use of synthetic absorptive matrices (SAM) for detection of respiratory pathogens versus nasopharyngeal swabs (NPS) and saliva; Assess dynamics of URT infection/colonisation and examine its relationship with symptoms, host responses and microbiota; Measure transmission between children and parents and immune responses in parents.

Study design: Prospective community-based cohort study.total of 45 children, aged 1-5 years old attending daycare or (pre-)school, will be included, including a pilot of 10 children to assess tolerability. If there are insufficient pneumococcal acquisitions in the study to assess the primary outcome, additional children can be recruited in groups of 3 or 4 children (up to 10). For a subset of participating children, both parents will be asked to self-collect daily saliva during the study.

Primary study parameters: Frequency of systemic polysaccharide specific B cells in children that become colonised during the study versus children that do not become colonised Secondary study parameters: Dynamics of respiratory bacteria and viruses during URT infection/colonisation. Presence and load for bacteria and viruses in children in SAM versus saliva and NPS. Local microbiota and immune profiles and association with infection/colonisation and symptomology. For a subset of parents, daily presence and load of bacteria and viruses as well as host immune factors measured in saliva.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from all legal representatives, for example both parents.
* Child aged 1-5 years of age attending day care, peuterspeelzaal or school at least 2 (half) days a week.
* Parents ability and willingness to adhere to protocol-specified procedures, including availability of a freezer at home to store samples. This does not include donation of saliva by parents themselves, which is related to a secondary endpoint.

Exclusion Criteria:

* History of respiratory tract infections requiring hospitalization
* Current use of antibiotics, or antibiotics use in past four weeks
* Use of immune-altering medication (such as steroids, including inhaled corticosteroid)
* No history of severe concomitant disease (severe congenital heart disease, bronchopulmonary dysplasia, prematurity <32 weeks, cystic fibrosis, sickle cell disease, congenital or acquired immunodeficiency disorders, cardiovascular disease, neuromuscular disorders, oncology patients or major congenital anomalies)

Ages: 1 Year to 5 Years | Sex: All
Age Groups: Child
Study Population: Children aged 1-6 years old, as these are a main population at risk for severe respiratory tract infections, and a main source of transmission. The study team will recruit families from the area of North/South-Holland as this will facilitate the home visits.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Frequency of systemic polysaccharide specific B cells in children that become colonised during the study versus children that do not become colonised | up to study completion, 28 or 29 days

SECONDARY OUTCOMES:
The number of participants with pneumococcal colonisation presence over time. | up to study completion, 28 or 29 days
  lyta, piab and serotype-specific qPCR
Pneumococcal colonisation density over time. | up to study completion, 28 or 29 days
  lyta, piab and serotype-specific qPCR
The number of participants with presence of other bacteria and viruses | up to study completion, 28 or 29 days
  Presence of other respiratory bacteria (such as Haemophilus influenzae and Staphylococcus aureus) and viruses (such as coronaviruses and influenza virus) during URT infection/colonisation, measured by molecular methods.
Density of other bacteria and viruses | up to study completion, 28 or 29 days
  Density of other respiratory bacteria (such as Haemophilus influenzae and Staphylococcus aureus) and viruses (such as coronaviruses and influenza virus) during URT infection/colonisation, measured by molecular methods.
Local microbiome composition measured by 16S | up to study completion, 28 or 29 days
  Relative abundance of ASV
Nasal and systemic antibodies titres specific for identified pathogens, measured using ELISA or antigen arrays | up to study completion, 28 or 29 days
  antigen-specific IgG, IgA and IgM titres
Nasal cytokine levels, assessed using multiplex assays such as Luminex | up to study completion, 28 or 29 days
  Individual cytokines will be reported in absolute or relative values
Symptom questionnaires | up to study completion, 28 or 29 days
  Symptoms are scaled on presence/absence
Evaluation/Sample tolerability questionnaires | day 28, last visit
  scale includes completely disagree, disagree, neutral, agree, completely agree for each question
Presence of bacteria and viruses in saliva of a subset of parents on a daily interval | up to study completion, 28 or 29 days
  Measured using molecular methods
Density of bacteria and viruses in saliva of a subset of parents on a daily interval | up to study completion, 28 or 29 days
  Measured using molecular methods

CONTACTS AND LOCATIONS:
Overall Officials: Marlies A van Houten, MD, Principal Investigator — Spaarne Gasthuis
Locations (1):
- Spaarne Gasthuis, Hoofddorp, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
If any samples or data are shared to perform analyses as described in the study protocol, either inside or outside EU, only pseudonymized material is shared to ensure participant privacy.
  This can be done upon request and following the signing of MTA/DTA.
  Individual datasets might be placed on repositories with restricted access or fully anonymized (such as Zenodo or flowrepository.org) upon publication.